CLINICAL TRIAL: NCT02101801
Title: Urine Drug Levels Related to Source of Water for Irrigation for Vegetable Crops Among Healthy Israeli Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: orap2014-HMO-CTIL
Record Dates: First submitted 2014-02-27; First posted 2014-04-02 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2015-08

CONDITIONS: Healthy Individuals
Keywords: environment, recycled wastewater, carbamazepine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- freshwater (Other): receives vegetables from freshwater farms
  Interventions: Other: vegetables from fresh or recycled water; Other: receives vegetables from fresh water or recycled waste water farms
- recycled wastewater (Active Comparator): receives vegetables from farms using recycled wastewater irrigation
  Interventions: Other: vegetables from fresh or recycled water; Other: receives vegetables from fresh water or recycled waste water farms

INTERVENTIONS:
Other: vegetables from fresh or recycled water
Other: receives vegetables from fresh water or recycled waste water farms

SUMMARY:
Over 60% of crops in Israel are grown in recycled treated waste water. This study aims to determine whether minute quantities of drugs such as Carbamazepine can be found in individuals who ingest vegetables grown in waste water.

DETAILED DESCRIPTION:
40 healthy volunteers will undergo a food frequency questionnaire and ask to undergo a daily food diary.They will also be asked about drug exposure.

At baseline they will provide a urine and hair sample to determine presence of pharmaceuticals.

They will then undergo a crossover trial wih one week exposure to vegetables grown in recycled waste water or fresh water, with a three day wash out period. Participants will be asked to ingest a minimal amount of lettuce, carrots, peppers, tomatoes and lettuce during the study period.

During this period questionnaires will continue and urine samples will be collected every three days. The first compound to be tested will be carbamazepine, as it is stable in water.

It is important to note that vegetables provided to the participants are available in regular grocery stores.

Participants will be asked to drink bottled water throughout the study period . A sample of their home drinking water will also be tested for Carbamazepine as will a sample of the vegetables they consume.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age 18-68

Exclusion Criteria:

* ingestion of carbamazepine,
* pregnancy
* vegetarian
* pure organic diet

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2016-03-29 (Actual)

PRIMARY OUTCOMES:
mean urine carbamazepine level in parts per billion | two weeks
  Urine will be tested on days -3,0,4,8

CONTACTS AND LOCATIONS:
Overall Officials: Ora Paltiel, MDCM, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel